CLINICAL TRIAL: NCT04473703
Title: A Prospective Study of Cardiac Adverse Reactions Related to Immune Checkpoint Inhibitor in Non-Small Cell Lung Cancer Patients
Brief Title: Cardiac Adverse Reactions Related to Immune Checkpoint Inhibitor in NSCLC Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xumin Hou, Chief physician, Shanghai Chest Hospital
Other Study IDs: SHXKYY202005
Record Dates: First submitted 2020-07-14; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Adverse Reactions; Immune Checkpoint Inhibitor; Non-Small Cell Lung Cancer Patients; Cardiac Event
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observation group: A total of 300 patients are expected to include in this group. And the cardiac adverse reactions related to immune checkpoint inhibitor will be observed.
  Interventions: Drug: renin-angiotensin system inhibitors or angiotensin-receptor-neprilysin inhibitor

INTERVENTIONS:
Drug: renin-angiotensin system inhibitors or angiotensin-receptor-neprilysin inhibitor — Patients with odd random number will treat with RASI（renin-angiotensin system inhibitors）, and those with even random number will treat with ARNI（angiotensin-receptor-neprilysin inhibitor）

SUMMARY:
This is a prospective, open label, single arm study. A total of 300 patients with primary non-small cell lung cancer treated with PD-1/PD-L1 immune checkpoint inhibitors(ICIs) are expected to included . All patients will follow up for at least 1 year. Patients with cardiac adverse reactions after PD-1/PD-L1 immune checkpoint inhibitor treatment at admission or during the subsequently follow-up period will randomly assigned a random number to each patient by computer random sequence. Patients with odd random number will treat with RASI（renin-angiotensin system inhibitors）, and those with even random number will treat with ARNI（angiotensin-receptor-neprilysin inhibitor）.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial;
2. Lung cancer patients whose pathological results confirmed is primary non-small cell lung cancer, stage III~IV;
3. Patients received with ICIs treatment, including anti-PD-1 or anti-PD-L1 for at least two courses;

Exclusion Criteria:

1. Patients who do not have pathological diagnosis;
2. Patients who can't finish the follow-up;
3. The anti-PD-1, anti-PD-L1 therapy was less than two courses;
4. Patients whose cancer diagnosed with small cell lung cancer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 300 patients with primary non-small cell lung cancer treated with PD-1/PD-L1 immune checkpoint inhibitors(ICIs) are expected to included. And then the basic information and the examination results will be collected.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 1 year
  a) Primary Outcome is Major Adverse Cardiovascular Events（MACE）related to ICIs，includes: cardiovascular death, myocardial infarction(nonfatal), stroke(nonfatal), heart failure that caused readmission

SECONDARY OUTCOMES:
Common Terminology Criteria for Adverse Events (CTCAE) | 1 year
  Common Terminology Criteria for Adverse Events (CTCAE) related to ICIs, includes: arrhythmia, cardiogenic chest pain, valvular heart disease, cardiomyopathy, myocardial pericardial disease
All cause of death | 1 year
  every reason that cause patient's death after ICIs treatment
examination indexes | 1 year
  The examination indexes that related to myocardial damage

IPD SHARING:
Plan to Share IPD: Undecided